CLINICAL TRIAL: NCT01825460
Title: Short-Term Effects of a Manual Therapy Protocol
Brief Title: Manual Therapy to Treat Acute Whiplash Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Universidad de Granada (Other); Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD (Lecturer), Universidad de Almeria
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UAL-326
Record Dates: First submitted 2013-03-27; First posted 2013-04-05 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-05

CONDITIONS: Whiplash Injuries
Keywords: Cervical spine; Neck pain; Manual therapy; Controlled clinical trial
MeSH Terms: conditions — Whiplash Injuries; Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Therapy Protocol (Experimental): A protocol with five techniques on thoracic area applied twice a week.
  Interventions: Other: Manual Therapy Protocol
- Two manual techniques (Active Comparator): Two manual therapies on thoracic area applied twice a week.
  Interventions: Other: Two manual techniques

INTERVENTIONS:
Other: Manual Therapy Protocol — The manual therapy protocol consists in the application of the following techniques: stretching diaphragm, Inhibition for phrenic center, Neuromuscular technique, technique jones and balance technique functional.
  Arms: Manual Therapy Protocol
Other: Two manual techniques — The two manual techniques applied to control group are: inhibition for phrenic center and neuromuscular technique.
  Arms: Two manual techniques

SUMMARY:
The purpose of this study is to determine the short-term effects of a manual therapy protocol on pain, disability and cervical range of motion in individuals with acute whiplash injury.

DETAILED DESCRIPTION:
Design: Randomized clinical trial. Objectives: to determine the short-term effects of a a manual therapy protocol on pain, disability and cervical range of motion in individuals with acute whiplash injury.

Methods and measures: sixty patients will be randomly assigned to 1 of 2 groups: the experimental group received a manual therapy protocol and the placebo group received two manual therapy techniques. Neck pain, disability and cervical range of motion data will be collected at baseline and 24-hr after the last manual therapy application. Mixed-model analyses of variance will be used to examine the effects of the treatment on each outcome variable.

ELIGIBILITY:
Inclusion Criteria:

* To met Quebec Task Force Classification of WAD II- neck pain symptoms and musculoskeletal signs.
* No evidence of conduction loss on clinical neurological examination.

Exclusion Criteria:

* Concussion during the motor vehicle accident.
* Loss of consciousness.
* Head or upper quadrant injury during the accident.
* Sought treatment prior to their accident for neck pain.
* A previous history of whiplash
* Neck pain
* Headaches
* Psychiatric or psychologic condition
* Neurologic or circulatory disorders

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change on Numerical Pain Rating Scale | At baseline and 2 weeks
  The numerical pain rating scale is used to record the patient´s current level of neck pain.

SECONDARY OUTCOMES:
Neck disability index | At baseline and 2 weeks
  The neck disability index consists of 10 questions addressing functional activities such as personal care, lifting, reading, work, driving, sleeping, recreational, pain intensity, concentration and headache.
Cervical Range of Motion | At baseline and 2 weeks
  Cervical range of motion is assessed with the patient sitting comfortably on a chair, with both feet flat on the floor, hips and knees at 90º of flexion, and buttocks positioned against the back of the chair.
Tampa scale for kinesiophobia | At baseline and 2 weeks
  The 17-item Tampa scale for kinesiophobia assesses fear of movement or of injury or reinjury.

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida M Castro-Sánchez, PhD, Study Director — Universidad de Almeria
Locations (1):
- Adelaida María Castro-Sánchez, Almería, Almeria, Spain

REFERENCES:
- [Background] Elliott JM, Kerry R, Flynn T, Parrish TB. Content not quantity is a better measure of muscle degeneration in whiplash. Man Ther. 2013 Dec;18(6):578-82. doi: 10.1016/j.math.2013.02.002. Epub 2013 Mar 5. PMID 23465963
- [Background] Smith J, Bolton PS. What are the clinical criteria justifying spinal manipulative therapy for neck pain?- a systematic review of randomized controlled trials. Pain Med. 2013 Apr;14(4):460-8. doi: 10.1111/pme.12041. Epub 2013 Feb 22. PMID 23432939
- [Background] Humphreys BK, Peterson C. Comparison of outcomes in neck pain patients with and without dizziness undergoing chiropractic treatment: a prospective cohort study with 6 month follow-up. Chiropr Man Therap. 2013 Jan 7;21(1):3. doi: 10.1186/2045-709X-21-3. PMID 23295018
- [Background] Isabel de-la-Llave-Rincon A, Puentedura EJ, Fernandez-de-Las-Penas C. Clinical presentation and manual therapy for upper quadrant musculoskeletal conditions. J Man Manip Ther. 2011 Nov;19(4):201-11. doi: 10.1179/106698111X13129729551985. PMID 23115473
- [Background] Pedler A, Motlagh H, Sterling M. Laterality judgments are not impaired in patients with chronic whiplash associated disorders. Man Ther. 2013 Feb;18(1):72-6. doi: 10.1016/j.math.2012.07.006. Epub 2012 Sep 5. PMID 22959229
- [Background] Stone AM, Vicenzino B, Lim EC, Sterling M. Measures of central hyperexcitability in chronic whiplash associated disorder--a systematic review and meta-analysis. Man Ther. 2013 Apr;18(2):111-7. doi: 10.1016/j.math.2012.07.009. Epub 2012 Sep 1. PMID 22947552
- [Background] Goldsmith R, Wright C, Bell SF, Rushton A. Cold hyperalgesia as a prognostic factor in whiplash associated disorders: a systematic review. Man Ther. 2012 Oct;17(5):402-10. doi: 10.1016/j.math.2012.02.014. Epub 2012 Mar 29. PMID 22464187
- [Background] Oddsdottir GL, Kristjansson E. Two different courses of impaired cervical kinaesthesia following a whiplash injury. A one-year prospective study. Man Ther. 2012 Feb;17(1):60-5. doi: 10.1016/j.math.2011.08.009. Epub 2011 Sep 28. PMID 21955671
- [Background] Picelli A, Ledro G, Turrina A, Stecco C, Santilli V, Smania N. Effects of myofascial technique in patients with subacute whiplash associated disorders: a pilot study. Eur J Phys Rehabil Med. 2011 Dec;47(4):561-8. Epub 2011 Jul 28. PMID 21796089
- [Background] Verhagen AP, Lewis M, Schellingerhout JM, Heymans MW, Dziedzic K, de Vet HC, Koes BW. Do whiplash patients differ from other patients with non-specific neck pain regarding pain, function or prognosis? Man Ther. 2011 Oct;16(5):456-62. doi: 10.1016/j.math.2011.02.009. Epub 2011 Mar 13. PMID 21406332
- [Background] Stokell R, Yu A, Williams K, Treleaven J. Dynamic and functional balance tasks in subjects with persistent whiplash: a pilot trial. Man Ther. 2011 Aug;16(4):394-8. doi: 10.1016/j.math.2011.01.012. Epub 2011 Mar 1. PMID 21367648
- [Background] Johansson MP, Baann Liane MS, Bendix T, Kasch H, Kongsted A. Does cervical kyphosis relate to symptoms following whiplash injury? Man Ther. 2011 Aug;16(4):378-83. doi: 10.1016/j.math.2011.01.004. Epub 2011 Feb 3. PMID 21295511
- [Background] Yu LJ, Stokell R, Treleaven J. The effect of neck torsion on postural stability in subjects with persistent whiplash. Man Ther. 2011 Aug;16(4):339-43. doi: 10.1016/j.math.2010.12.006. Epub 2011 Jan 20. PMID 21256074